CLINICAL TRIAL: NCT00347568
Title: BC-DAISY: A Breast Cancer Decision Aid System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0312-05
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: decision aids; high risk; breast cancer; breast cancer prevention
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Device: TX-plore — PI has terminated at institution and there is no one available to report.

SUMMARY:
The purpose of this study is to develop a web-based decision aid to help women at high risk for breast cancer make informed breast cancer prevention choices. These choices include chemoprevention, surgery, genetic counseling, or regular screening in accordance with recommended guidelines.

DETAILED DESCRIPTION:
Decisions about breast cancer are complex and preference-based. Existing decision aids that help identify women eligible for tamoxifen based on their breast cancer risk, such as the Breast Cancer Risk Assessment Tool (BCRAT), were not designed to identify women's risks for side-effects, her preferences for outcomes affected by treatment, nor the net balance of benefits and risks. It is possible to predict the risks of side effects of treatments according to patient characteristics, using patient-specific models.Our goal is to develop a decision aid, TXplore, that rates the overall benefit:risk profiles of various breast cancer prevention strategies according to a woman's risks for breast cancer, side-effects, and preferences. Each user will receive a customized report card grading each available prevention option, using preference-weighted risk:benefit grades; users can also explore personalized feedback from the program. Our hypotheses are that this tool can improve the implementation of appropriate prevention strategies, promote risk reduction behavior, and improve PCP's ability to identify and counsel high risk women.We propose building on modeling techniques that link the benefits and risks of preventive strategies to patient characteristics and preferences. We now seek to conduct focus groups and usability tests on end-users to optimize the design of the prototype TXplore.

The Specific Aims are:

1. To optimize the design of TXplore by focus groups conducted among diverse high-risk women and PCPs to a) identify the domains driving decisions about prevention and explore the framing of questions comparing the relative importance of one domain to another, synthesizing this information as preference trade-off questions; and b) explore the framing of risk:benefit grades and personalized feedback.
2. To assess the comprehensibility of preference trade-off questions by testing each question on a diverse sample of 50 high-risk women, revising and retesting.
3. To assess the usability of TXplore for patients and PCPsThe successful completion of this project will produce a novel tool for counseling women about their individual benefits and risks of breast cancer prevention strategies. It will be the first tool of its kind to integrate individual patient risks and preferences into decision support.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 21 - 75
* at least one first degree relative with breast cancer or a Gail Model score signifying high risk
* female
* having had contact with a PCP (physician or nurse practitioner)within the last year
* being a patient at a participating clinic (for usability and pilot study)

Exclusion Criteria:

* Inability to give informed, voluntary consent
* History of breast cancer or LCIS
* Language, vision, or reading difficulties, or non-English speaking
* Pregnancy
* women over 75 because of the lack of data guiding the impact of preventive treatments among this age group.

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Usability feedback on new decision aid for women at high risk for breast cancer from patients and physicians. | 9/01/06-8/31/07

CONTACTS AND LOCATIONS:
Overall Officials: Nananda Col, MD, MPP, MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States